CLINICAL TRIAL: NCT00370253
Title: Noradrenalin vs Terlipressin in Patients With Hepatorenal Syndrome.A Prospective, Randomized Study
Brief Title: Noradrenalin vs Terlipressin in Hepatorenal Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Mario Rizzetto, University of Turin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA-TER
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Hepatorenal Syndrome
Keywords: hepatorenal syndrome; ascites; portal hypertension; cirrhosis
MeSH Terms: conditions — Hepatorenal Syndrome; Ascites; Hypertension, Portal; Fibrosis | interventions — Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Terlipressin
  Interventions: Drug: Terlipressin
- 1 (Experimental): Noradrenalin
  Interventions: Drug: Noradrenalin

INTERVENTIONS:
Drug: Terlipressin — 1mg/4 h per day
  Arms: 2
Drug: Noradrenalin — 0,1 mcg/kg/min
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether noradrenalin is as effective and safe as terlipressin in the treatment of hepatorenal syndrome

DETAILED DESCRIPTION:
Hepatorenal syndrome (HRS) is a major complication of cirrhosis; it is characterized by functional renal failure and poor prognosis. Arterial dilation is a key pathogenic event of HRS, leading to reduction of the effective blood volume, homeostatic activation of vasoactive systems and renal vasoconstriction with decrease in renal blood flow. The clinical signs of HRS vary depending on the clinical pattern. HRS type 1 is characterized by a rapidly progressive renal failure; HRS type 2 by a moderate and more stable renal failure. HRS type 1 has a very poor short term prognosis, with a median survival of only about 2 weeks; patients with HRS type 2 have a median survival of about 6 months. The management of HRS still constitutes a major challenge. Liver transplantation is the ideal treatment, but it has important inherent drawbacks, such as the organ shortage and the time needed to perform the transplant, that is too long to consent the survival of these patients. The management of HRS has focused on improving renal function, thus extending patients survival and allowing the performance of the liver transplant. In the last years, remarkable results have been obtained using vasoconstrictor drugs. By improving the effective blood volume, vasoconstrictors induce the suppression of homeostatic vasoactive systems and increase renal blood flow and glomerular filtration rate.Among vasoconstrictors, terlipressin, a V1 vasopressin agonist, has currently the best efficacy pedigree. However, it is expensive and is not available in many countries, including North America. More recently, it was suggested that alpha-adrenergic drugs such noradrenalin and midodrine may be also effective in HRS. Noradrenalin would have the potential advantage of wider availability and of lower cost. The current prospective randomized study was undertaken to assess the efficacy and safety of noradrenalin vs terlipressin in patients with HRS.

ELIGIBILITY:
Inclusion Criteria:

* Hepatorenal syndrome
* Age: 18-75 years
* Informed written consent

Exclusion Criteria:

* Multinodular hepatocellular carcinoma (more than 3 nodules)
* Portal vein thrombosis
* Ongoing bacterial infection
* Ongoing or recent (less than one week) bleeding
* Cardio-pulmonary failure
* Coronary artery disease
* Peripheral artery disease
* Arterial hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Renal function at the beginning and at the end of therapy | two weeks

SECONDARY OUTCOMES:
Circulatory function | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mario Rizzetto, MD, Study Director — Division of Gastroenterology and Hepatology, San Giovanni Battista Hospital, Turin, Italy
Locations (1):
- San Giovanni Battista Hospital, Turin, Italy

REFERENCES:
- [Background] Ortega R, Gines P, Uriz J, Cardenas A, Calahorra B, De Las Heras D, Guevara M, Bataller R, Jimenez W, Arroyo V, Rodes J. Terlipressin therapy with and without albumin for patients with hepatorenal syndrome: results of a prospective, nonrandomized study. Hepatology. 2002 Oct;36(4 Pt 1):941-8. doi: 10.1053/jhep.2002.35819. PMID 12297842
- [Background] Duvoux C, Zanditenas D, Hezode C, Chauvat A, Monin JL, Roudot-Thoraval F, Mallat A, Dhumeaux D. Effects of noradrenalin and albumin in patients with type I hepatorenal syndrome: a pilot study. Hepatology. 2002 Aug;36(2):374-80. doi: 10.1053/jhep.2002.34343. PMID 12143045
- [Derived] Alessandria C, Ottobrelli A, Debernardi-Venon W, Todros L, Cerenzia MT, Martini S, Balzola F, Morgando A, Rizzetto M, Marzano A. Noradrenalin vs terlipressin in patients with hepatorenal syndrome: a prospective, randomized, unblinded, pilot study. J Hepatol. 2007 Oct;47(4):499-505. doi: 10.1016/j.jhep.2007.04.010. Epub 2007 May 24. PMID 17560680